CLINICAL TRIAL: NCT04810182
Title: Regorafenib in Relapsed Glioblastoma. An Observational, Multicentric and Prospective Study. IOV-GB-1-2020 REGOMA-OSS
Brief Title: Regorafenib in Patients With Relapsed Glioblastoma. IOV-GB-1-2020 REGOMA-OSS
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IOV-GB-1-2020 REGOMA-OSS
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — regorafenib; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glioblastoma Patients treated with Regorafenib: Patients with a confirmed diagnosis of Glioblastoma for whom a decision to treat with regorafenib has been made (by the treating physician).
  Interventions: Drug: Regorafenib 40 MG Oral Tablet [STIVARGA]

INTERVENTIONS:
Drug: Regorafenib 40 MG Oral Tablet [STIVARGA] — As per the treating physicians discretion

SUMMARY:
This study aims to analyze the role the of Regorafenib in prolonging the Overall Survival of glioblastoma multiforme patients who progressed after surgery and a first-line chemo-radiotherapy treatment in the setting of "real world life".

DETAILED DESCRIPTION:
The primary aim of the study

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Histologically confirmed glioblastoma (grade IV)
* First recurrence after adjuvant treatment (surgery followed by radiotherapy and temozolomide chemotherapy) in patients who have not received further therapeutic interventions
* World Health Organization (WHO) Performance status ≤ 1 (or Karnofsky performance status (KPS) ≥70)) before the start of the treatment
* Documented progression of disease as defined by RANO criteria at least 12 weeks after completion of radiotherapy, unless the recurrence is outside the radiation field or has been histologically documented.
* Documented progression of disease by a brain MRI scan done within 14 days before the start of treatment with Regorafenib.
* Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
* Have adequate bone marrow function, liver function, and renal function, as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:
* Hemoglobin >9.0 g/dl
* Absolute neutrophil count (ANC) >1500/mm3 without transfusions or granulocyte colony stimulating factor and other hematopoietic growth factors
* Platelet count ≥100,000/μl
* White blood cell count (WBC) >3.0 x 109/L
* Total bilirubin <1.5 times the upper limit of normal
* ALT and AST <3 x upper limit of normal
* Serum creatinine <1.5 x upper limit of normal
* Alkaline phosphatase <2.5 x ULN (<5 x upper limit of normal value)
* PT-INR/PTT <1.5 x upper limit of normal
* Lipase ≤ 1.5 x the ULN
* Glomerular filtration rate ≥ 30 mL/min/1.73 m2
* TSH, fT3,fT4 within normal limits
* Patients may have undergone surgery for the recurrence; the histological report must document a glioblastoma recurrence. If operated:
* at least 28 days from the surgery is required prior to Regorafenib administration and patients should have fully recovered.

Exclusion Criteria:

* Have had prior treatment with regorafenib or any other VEGFR-targeting kinase inhibitor
* Have had systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and/or hormonal therapy within 4 weeks prior to initiation of treatment
* Recurrent disease located outside of the brain
* Have uncontrolled hypertension (systolic blood pressure [SBP] > 140 mmHg or diastolic blood pressure [DBP] > 90 mmHg) despite optimal medical management
* Have had a myocardial infarction < 6 months prior to initiation of treatment with Regorafenib
* Have had arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months prior to the initiation of treatment with Regorafenib
* Have either active or chronic hepatitis B or C requiring treatment with antiviral therapy
* Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapse of glioblastoma (grade IV) after surgery and radio-chemotherapy first line treatment, treated with Regorafenib until disease progression or the appearance of unacceptable toxicity.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the enrolment date to the date of death, for any cause, or to the last follow-up, assessed up to 18 months
  Overall Survival is defined as the time from date of enrolment to the date of death due to any cause

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the date of enrolment to the date of disease progression or to the date of death, assessed up to 18 months
  from the date of enrolment to the date of disease progression determined using RANO criteria or to the date of death, whichever occurs first.
Objective response rate (ORR) | Approximately 24 months
  As percentage of patients achieving a complete response plus partial response
Disease control rate (DCR) | Approximately 24 months
  As percentage of patients achieving a complete response plus partial response plus stable disease.
Toxicity (Graded according to the NCI-Common Terminology Criteria for Adverse Events-CTCAE v5.0) | From the start of Regorafenib treatment up to 30 days after the end of treatment
  Toxicity during the treatment will be recorded and graded according to the NCICommon Terminology Criteria for Adverse Events (CTCAE) v.4.. , related to severity of the adverse event from Grade 1 to Grade 5

CONTACTS AND LOCATIONS:
Locations (29):
- Italy (29):
  - Ospedale Generale Regionale " F.Miulli ", Acquaviva delle Fonti, BA
  - Policlinico Universitario di Bari, Bari, BA
  - IRCCS "Saverio de Bellis", Castellana Grotte, BA
  - Ospedlae S. Martino, Belluno, BL
  - Ospedale Bellaria, Bologna, BO
  - Ospedale Perrino, Brindisi, BR
  - Università e ASST Spedali Civili, Brescia, BS
  - Irst-Irccs, Meldola, FC
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, FI
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Ospedale Civile di Livorno, Livorno, LO
  - Ospedale Generale Provinciale, Macerata, MC
  - AOU Policlinico "G.Martino", Messina, ME
  - Istituto Neurologico C. Besta IRCCS, Milan, MI
  - Ospedale Humanitas, Rozzano, MI
  - Ospedale del Mare, Napoli, NL
  - Fondazione Istiuto Giglio Cefalù, Cefalù, PA
  - Aulss6 Euganea Padova Sud Ospedali Riuniti, Piove di Sacco, PD
  - Azienda Ospedaliero Universitaria di Pisa, Pisa, PI
  - Istituto Nazionale Tumori Regina Elena -IFO, Roma, RM
  - Policlinico Universitario Gemelli, Roma, RM
  - Ospedale di Rovigo, Rovigo, RO
  - Azienda Ospedaliero Universitaria di Siena, Siena, SI
  - Azienda Ospedaliero Universitaria della Città della Salute e della Scienza, Torino, TO
  - Azienda Ospedaliera Santa Maria, Terni, TR
  - Ospedale San Donà di Piave _Azienda ULSS 4 " Veneto Orientale", San Donà di Piave, VE
  - AULSS 7 Distretto 2 Ospedale Santorso, Santorso, VI
  - AULSS 9 Scaligera Ospedale Mater Salutis, Legnago, VR
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine